CLINICAL TRIAL: NCT06877403
Title: Prospective Study on the Prevalence and Impact of Fatigue in Myasthenic Patients Followed At Clermont-Ferrand University Hospital - "My" Asthenia
Brief Title: Prevalence and Impact of Fatigue in Myasthenic Patients Followed At Clermont-Ferrand University Hospital - "My" Asthenia
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 TAITHE
Record Dates: First submitted 2025-02-25; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Myasthenia Gravis
Keywords: observationnal; fatigue; self-questionnaires; myasthenia gravis; ocular myasthenia gravis; generalized myasthenia gravis; comorbidities
MeSH Terms: conditions — Myasthenia Gravis; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients suffering from myasthenia gravis (MGFA I to IV) followed in Clermont-Ferrand: Adult patients who consulted the neurology department of the Clermont-Ferrand University Hospital between 01/01/2022 and 12/31/2024 in the context of their myasthenia and identified by the BAMARA and PMSI databases of the Clermont-Ferrand University Hospital Diagnosis of autoimmune myasthenia gravis based on biological and/or electromyographic criteria MGFA class from I to IV

SUMMARY:
After identifying myasthenic patients meeting the inclusion criteria, telephone contact with patients to suggest that they participate in the study by responding to various questionnaires composed of validated scales used in current practice (MG-ADL, MG-QoL-15, MFIS, FSS, PASS, HADS, Godin-Leisure Exercise Time) which will be completed either digitally (REDCap link) or by paper form if necessary. Consultation of patients' medical records to collect information relating to factors associated with fatigue or intrinsic illness (demographic data, comorbidities, progression of the illness, treatments, etc.).

As part of their usual care, myasthenia patients answer questionnaires according to the following procedure :

1. Mailing of questionnaires to all eligible patients before their consultation The questionnaires are composed of scales validated and used in current practice (MG-ADL, MG-QoL-15, MFIS, FSS, PASS, HADS, Godin-Leisure Exercise Time).
2. Collection of questionnaires When patients come for consultation, the completed questionnaires are collected by the medical team.
3. Collection of questionnaires The responses to the questionnaires and the scores and results obtained from these questionnaires are integrated into the patients' medical records.

As part of our study and in parallel with the patient's clinical follow-up, data relating to factors associated with fatigue or intrinsic illness (demographic data, comorbidities, progression of the disease, treatments, etc.) as well as responses to questionnaires will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who consulted the neurology department of the Clermont-Ferrand University Hospital between 01/01/2022 and 12/31/2024 in the context of their myasthenia and identified by the BAMARA and PMSI databases of the Clermont-Ferrand University Hospital
* Diagnosis of autoimmune myasthenia gravis based on biological and/or electromyographic criteria
* MGFA class from I to IV

Exclusion Criteria:

* Patients under guardianship or curatorship
* Non-French speaking patients
* Patients refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Myasthenic patients with ocular or generalized form followed in Clermont Ferrand University Hospital (MGFA I to IV)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of fatigue | through study completion, an average of 6 month
  Determine the prevalence of fatigue in myasthenic patients followed at the Clermont-Ferrand University Hospital by the Fatigue Severity Scale from 1 to 7. 1 = not significative fatigue. 7 = extreme fatigue. Significant if FSS > 4.

SECONDARY OUTCOMES:
Impact of the fatigue | through study completion, an average of 6 month
  Describe the impact of fatigue on daily life by the Modified Fatigue Impact Scale from 21 to 84. 21 = not significative impact of fatigue on daily life, 84 = severe impact of the fatigue. Significant if MFIS > 45.

OTHER OUTCOMES:
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Disease severity by MG-ADL (from 0 to 24), 0 means no symptom, 24 means severe symptoms. No specific threshold.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Impact of the disease on the daily-life activities by the MG-QoL-15 (from 0 to 60), 0 means no repercussion, 60 means massive repercussion. No specific threshold.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Level of anxiety and depression by HADS (< 7 : no symptoms, 8 -11 doubt, > 11 symptoms of anxiety and depression)
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. level of physical activity by Godin Leisure Time Activity Questionnaire (> 24 : active, 14-23 moderate activity, < 14 sedentary)
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Global feeling about the myasthenia by a simple question with the PASS (yes / no)
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic : age in years.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic : weight in kilograms, height in meters, BMI in kg/m2
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic : duration of the disease in years
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic : type of actual or passed treatment : corticoids, anticholinesterasic, immunosuppressive (Azathioprine, Mycophenolate mofetil, Ciclosporine, Rituximab), novel therapy (Efgartigimod-alpha, Zilucoplan, Ravulizumab). Yes or No for each treatment.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic : dosage of actual or passed treatment (corticoids, anticholinesterasic, immunosuppressive (Azathioprine, Mycophenolate mofetil, Ciclosporine, Rituximab), novel therapy (Efgartigimod-alpha, Zilucoplan, Ravulizumab). Dosage in mg per day
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic and notably comorbidities : auto-immune (dysthyroiditis, diabete, lupus, rheumatoid arthritis, other). Yes or No.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic and notably comorbidities : thymectomy. Yes or No.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic and notably comorbidities : date of the last myasthenic crisis. Month and years or the year exclusively.
Associated factors with fatigue | through study completion, an average of 6 month
  Study the factors associated with fatigue. Analysis of the medical record for demographic and notably comorbidities : date of the last use of crisis treatment (Immunoglobulin, Plasmatic Exchange). Date in month and years or the year exclusively.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Taithe, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France